CLINICAL TRIAL: NCT04781907
Title: Patient Performed Tissue Expansion for Two-stage Alloplastic Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Research Priorities
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1704; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); UW20171 (Other: UWCCC); Protocol Version 2/25/2021 (Other: UW Madison)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Tissue Expansion; Breast Reconstruction
MeSH Terms: interventions — Tissue Expansion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Expansion Group (Experimental): Participants in home expansion group will perform the saline injection for their right tissue expander under clinic staff supervision on their 2nd and 3rd expansion. Beginning their 4th expansion, participants will perform saline injection at home prior to their regularly scheduled clinic visit.
  Interventions: Procedure: Tissue Expansion
- Control Group (No Intervention): Standard of Care

INTERVENTIONS:
Procedure: Tissue Expansion — Tissue expanders are used to increase the soft tissue envelope after mastectomy to provide adequate and healthy coverage of prosthetic breast implants.
  Arms: Home Expansion Group

SUMMARY:
This study is designed to evaluate the feasibility and safety of patient performed tissue expansions in two-stage alloplastic breast reconstruction with tissue expanders. The investigators hypothesize that a motivated patient who learns and demonstrates proper technique can safely perform tissue expansions at home, with no increase in complications or problems with reconstruction. 30 participants will be recruited for this study, 10 into a Home Expansion Group, and 20 into a Control Group.

DETAILED DESCRIPTION:
Two-stage tissue expander-to-implant reconstruction is the most common technique for breast reconstruction in the United States. Tissue expanders are used to increase the soft tissue envelope after mastectomy to provide adequate and healthy coverage of prosthetic breast implants. The current clinical standard of care entails an initial surgery for the placement of tissue expander device either in front or behind of the pectoralis muscle following a mastectomy. After an interval of a few weeks to allow surgical wound healing, the patient will make serial office visits (usually weekly) where the plastic surgeon or other clinical staff will inject the device with a bolus of saline. A probe is used to find the magnetic port embedded in the expander, which is then accessed with a sterile butterfly needle connected to a large syringe filled with saline. The serial injections continue until the tissue expander(s) have reached the desired size. The patient then undergoes a second surgery about 4-6 weeks after the last injection, to exchange the tissue expander with a breast implant.

The tissue expansion process can be inconvenient for the patient, due to the time and cost associated with travel and coordination of frequent office visits. The office visits for tissue expander injections ultimately result with multiple additional encounters with a healthcare facility, which may be of concern to patients, in light of the COVID-19 pandemic.

The saline tissue expander with internal filling port is still the clinical gold standard device for alloplastic breast reconstruction. But the safety, time benefits and healthcare utilization and cost savings of home inflation - as shown in studies using external filling port tissue expanders and carbon dioxide-filled tissue expanders - suggests that patient performed tissue expansions may also be feasible with conventional saline tissue expanders. This would obviate multiple outpatient visits usually required for saline injections. Eliminating the need for saline injection clinic visits would benefit both the clinician and patient/families by reducing financial and time burdens, and limit potential exposures to COVID-19.

Study Design:

Ten women age 18 or above who met the inclusion and exclusion criteria below will be recruited and enrolled in the study. Study participants will be recruited from the principal investigator's clinic. Surgical technique and timing for initiation of expansion and implant exchange will be performed according to the principal investigator's usual protocol with saline tissue expanders. At the first expansion clinic visit, the saline injection will be performed by clinic staff, as per usual protocol. Clinic staff will provide teaching on the saline injection technique during this visit. At the second and third clinic visit, the participant will perform the saline injection under supervision by clinic staff in the right breast, the left breast will be expanded by the clinic staff. Starting the fourth expansion, participants will perform expansion in right breast prior to their clinic visit and left breast will be expanded by clinic staff. Thus participants will still be seen in person on a regular basis as per usual clinical protocol. If after the second and third visit the participant is unable to demonstrate ability and comfort to perform expansions on her own after the third clinic visit, she will be excluded from the study. Participants will be provided instructional materials and all supplies necessary to perform expansions at home. After the tissue expanders have been fully expanded, the participant will proceed to undergo the principal investigator's usual protocol of exchange to breast implants.

If at any time the participant has problem with home expansion or no longer wants to be part of the study, she can leave the study and receive all expansions in the clinic per usual protocol.

Objectives:

* 1. Evaluate overall treatment success in undergoing alloplastic breast reconstruction
* 2. Evaluate profile and rate of complications in patients performing tissue expansions at home
* 3. Compare treatment success and complication profile/rate of right (patient performed tissue expansion) and left (clinic performed tissue expansion) breast
* 4. Compare treatment success and complication profile/rate of patients who perform some tissue expansions at home vs patients who have all tissue expansions performed by clinical staff
* 5. Evaluate patient's satisfaction in experience of learning and performing expansions at home

ELIGIBILITY:
Inclusion Criteria:

* Undergoing two stage bilateral alloplastic breast reconstruction with tissue expander (either immediate or delayed)
* Able and willing to present for clinic visits every 1-2 weeks per tissue expansion protocol
* Physical, perceptual and cognitive capacity to understand, learn, perform and manage at-home expansions
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Failure to demonstrate proper tissue expander saline infiltration technique after two teachings and observations by clinic staff
* Tissue integrity unsuitable for tissue expansion (compromised vascularity, history of compromised wound healing, mastectomy skin flaps of questionable viability, excessively tight skin envelope)
* Residual gross tumor at intended expansion site
* Current or prior infection at intended expansion site
* Clinically significant fibrosis caused by previous irradiation or planned radiation therapy at intended expansion site during time expander is implanted
* History of failed tissue expansion/breast implant reconstruction
* Concomitant medications that may place subject at increased risk of complications (adjuvant chemotherapy, therapeutic anticoagulation, steroids, immunosuppressants)
* Current tobacco smoker
* Comorbid condition that may place subject at increased risk of complications (severe collagen vascular disease, poorly managed diabetes, BMI > 35
* History of psychological condition, drug or alcohol misuse that may interfere with their ability to perform home expansions safely
* Participating in concurrent investigational drug or device study
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants who had their breast tissue expanders successfully exchanged from expander to implant | up to 6 months
  Clinically, the tissue expander is only temporary and the main goal is to get patient to their permanent breast implant
Incidence of Adverse Events | up to 6 months
  Adverse events including - wound dehiscence, seroma, hematoma, extrusion, capsular contracture

SECONDARY OUTCOMES:
Number of Right and Left breast tissue expanders successfully exchanged from expander to implant | up to 6 months
  Participants serve as internal control, with the right breast being expanded by self and left breast being expanded by clinical staff per usual protocol.
Incidence of Adverse Events in Left vs Right Breast Tissue Expansion | up to 6 months
  Participants serve as internal control, with the right breast being expanded by self and left breast being expanded by clinical staff per usual protocol.

OTHER OUTCOMES:
Participant Satisfaction Survey Score | up to 6 months
  Exit survey with 5-point Likert scale ratings on patient's experiences regarding tissue expansion process, where higher scores indicate increased satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Poore, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No